CLINICAL TRIAL: NCT02044718
Title: Medical Record Study on Adverse Events Requiring a Higher Level of Care in Flemish Hospitals
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); Algemeen Ziekenhuis Vesalius (Other); Sint-Franciscus Ziekenhuis (Unknown); Regionaal Ziekenhuis Sint-Trudo (Unknown); Ziekenhuis Maas en Kempen (Other); Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, prof. dr. Neree Claes, prof. dr., Hasselt University
Other Study IDs: 11.50/intens11.01
Record Dates: First submitted 2013-12-19; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Sepsis, Cancer, Heart Attack, Heart Failure, Abdominal Surgery, Trauma, Diabetes, Lung Disease, Gynaecology, Fertility, Cardiac Surgery,
Keywords: adverse events; unplanned admission intensive care; chart review
MeSH Terms: conditions — Sepsis; Neoplasms; Myocardial Infarction; Heart Failure; Wounds and Injuries; Diabetes Mellitus; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An adverse event (AE) is defined as unintended injury or complication, which results in disability, death or prolongation of hospital stay, and is caused by healthcare management (including omissions) rather than the patient's disease. Retrospective record reviews in several countries have shown that 2,9% to 16,6% of patients in acute hospitals experience one or more AEs. A patient with an AE may require a higher level of care. Although all AEs are important, preventable AEs that result in an upgraded level of patient care are of particular concern. In this study it's defined as an unplanned admission to intensive care unit (ICU) or a Mobile Emergency Team (MET) intervention. The objectives of this study are to determine the incidence of (preventable) adverse events requiring ICU admission or MET intervention and to assess the level of harm of each AE.

ELIGIBILITY:
Inclusion Criteria:

* All patients being transferred to a higher level of care during the study period (November 2011 - May 2012)
* In practice, the higher level of care means
* (1) (re)admission to the Intensive Care Unit from other care units in the hospital providing lower intensity care,
* (2) to an intervention by a Medical Emergency Team due to an unanticipated change in the patient's clinical status

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events requiring a higher level of care | 6 months
  An adverse event is an unintended injury or complication, which results in disability at discharge, death or prolongation of hospital stay, and is caused by healthcare management (including omissions) rather than the patient's disease. (Wilson, 1995)
The number of participants with preventable adverse events | 6 months
  Assess the preventability of these adverse events using six point scale with a range of not preventable until totally preventable

SECONDARY OUTCOMES:
Type adverse events | 6 months
  Divide the adverse events into categories, like diagnosis, therapy, medication, surgery, non-surgery, etc.
Clinical impact of adverse events in terms of outcome | 6 months
  Assess the impact of the adverse events in terms of disability, mortality, readmission.
Quality of the chart review | 6 months
  The patient chart will be judge on the completeness and adequacy

CONTACTS AND LOCATIONS:
Overall Officials: Kristel Marquet, drs, Principal Investigator — Hasselt University; Arthur Vleugels, prof. dr., Study Chair — KU Leuven
Locations (1):
- Hasselt University, Hasselt, Limburg, Belgium